CLINICAL TRIAL: NCT03736239
Title: Ultrasound Study of the Diaphragm Evolution Under ECMO
Acronym: DIAG-ECMO
Status: Completed | Type: Observational
Sponsor: Association Pro-arte (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2018-DIAGECMO
Record Dates: First submitted 2018-06-25; First posted 2018-11-09 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Cardiogenic Shock; Weaning Failure
Keywords: ECMO; Intensive Care Units; Shock, Cardiogenic; Ventilator Weaning; Diaphragm; Ultrasonography
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the evolution of diaphragmatic muscle effort in cardiogenic shock in ECMO patient with ultrasounds during the first weaning attempt in intensive care patients.

DETAILED DESCRIPTION:
Diaphragmatic atrophy and diaphragmatic dysfunction are described in human resuscitation under mechanical ventilation, but this diaphragmatic function has not been studied in patients with cardiogenic shock and also under cardiac assistance by extracorporeal circulation called ECLS (Extra -corporeal Life support). Diaphragmatic dysfunction in intensive care has been described during prolonged stay in intensive care and early sepsis. It is associated with dyspnea and delayed weaning from mechanical ventilation. The atrophy of the diaphragm muscle is related to both loss of function and also loss of muscle performance.

Decreases in heart muscle and diaphragm performance may require both cardiac and respiratory assistance. Cardiac and respiratory dysfunctions can complicate the weaning of the respiratory assistance and also extracorporeal circulatory support supports. These two supports, respiratory and circulatory assistance, allow the purification of CO2 and respiratory assistance is known to influence the diaphragmatic function. The role of the muscular pump function in the withdrawal process of the ECLS, remains largely unknown. The aim of our study is to give a description of the physiology of the diaphragm in case of cardiogenic shock: we want to evaluate the force of the diaphragm according to the ventilation under ECLS. No studies have yet evaluated the influence of ECLS as a CO2 purification system on the performance of the diaphragm muscle.

Ultrasound is used in the patient's bed in daily practice to measure cardiac function, vessel study and diaphragm muscle. This method is reproducible and non-invasive. It can be hypothesized that there is a muscular involvement of the diaphragm under extracorporeal membrane oxygenation (ECMO) measurable by ultrasound method. Our main hypothesis is that the diaphragm force evolves according to the cleaning of the CO2 by the ECLS during the weaning of this one.

This is a Monocentric Prospective Observational Descriptive study. The objective of this study is to evaluate prospectively and consecutively the evolution of diaphragmatic muscle stress in cardiogenic shock with ultrasounds during the first ECMO weaning in intensive care patients.

When cardiogenic shock occurs, during the first ECLS weaning, we also will evaluate prospectively :

* The evolution of diaphragm muscle thickness
* The evolution of the function of the diaphragm muscle We will evaluate the impact of different risk factors on the diaphragmatic function: respiratory variables, parameters and duration of mechanical ventilation, ECLS parameters and duration, number and type of associated organ failure, gasometric variables, hemodynamic variables, presence of a cardiotomy.

And we also will evaluate the impact of the diaphragmatic function on the patient's future:

* Failure to wean from mechanical ventilation
* ECLS weaning failure
* Death in intensive care
* Length of stay in intensive care Patients will be informed and consents will be collected during hospitalization in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care for cardiogenic shock under ECMO (extracorporeal membrane oxygenator)
* Veno-arterial ECMO
* ECMO withdrawal decision
* Patient or family agreeing to participate in research

Exclusion Criteria:

* Patient under guardianship or curatorship
* Contraindication to spontaneous ventilation
* Pregnant woman
* Anechoic patient for diaphragmatic ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited into the intensive care unit of the investigating center, under the responsibility of the principal investigator of the study. All patients admitted to intensive care present cardiogenic shock. After verification of the inclusion and non-inclusion criteria, the information on the diagnostic procedures will be given by one of the investigators.
  Due to the observational nature of the research, patients can participate in another one. There is not an exclusion period at the end of the search.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the evolution of the diaphragm muscle effort in cardiogenic shock during the first ECLS weaning in patients in ICU. | at 15 min
  The performance of the diaphragm muscle will be evaluated by ultrasonography (the thickening fraction of the diaphragm) during the weaning of the ECMO at different weaning level : after 15 minutes (Baseline, 4 l/min, 2 l / min, 1 l / min). Wash out of 10 min between each measurement. The parameters of the assisted ventilation will be standardized according to the practices of the service and recommendations.

SECONDARY OUTCOMES:
Evaluate prospectively during cardiogenic shock when weaning from ECLS, the evolution of diaphragm muscle thickness | at 15 min
  The thickness of the muscle will be measured when weaning the ECMO at the same scanning levels as before (mm).
Evaluate prospectively during cardiogenic shock when weaning from ECLS, the evolution of the function of the diaphragm muscle | at 15 min
  The function of the muscle will be measured when weaning the ECMO at the same scanning levels as before (%).
Evaluate the impact of different risk factors on the diaphragmatic function | previous exposure before inclusion
  Risk factors will be collected to estimate the impact on the 3 indicators of the diaphragm function (performance, thickness and function).
Evaluate the impact of the diaphragmatic function on the patient's future: failure to wean from mechanical ventilation | at 60 days
  Rate of weaning failure with mechanical ventilation will be collected
Evaluate the impact of the diaphragmatic function on the patient's future: ECLS weaning failure | at 60 days
  Rate of weaning failure with ECLS will be collected
Evaluate the impact of the diaphragmatic function on the patient's future: Death in intensive care | at 60 days
  Rate of mortality in intensive care will be collected.
Evaluate the impact of the diaphragmatic function on the patient's future: Length of stay in intensive care | at 60 days
  Length of stay in intensive care will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Henri Moury, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided
futur participation in respiratory protocols may include our datas.